CLINICAL TRIAL: NCT00790842
Title: A Phase I/II Study of the Tolerability of Lenalidomide and Low Dose Dexamethasone in Previously Treated Multiple Myeloma Patients With Impaired Renal Function
Brief Title: Lenalidomide and Low-Dose Dexamethasone in Patients With Previously Treated Multiple Myeloma and Kidney Dysfunction
Acronym: PrE1003
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: PrECOG, LLC. (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PrE1003; RV-MM-PrECOG-0394 (Other: Celgene Protocol)
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2018-10-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma; Plasma Cell Neoplasm
Keywords: Refractory Multiple Myeloma; Relapsed Multiple Myeloma; Multiple Myeloma with Renal Dysfunction; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Lenalidomide; Dexamethasone; Calcium Dobesilate; Anticoagulants; Aspirin; Heparin; Heparin, Low-Molecular-Weight; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group A - CrCl 30-60 mL/min (Experimental): Creatinine clearance 30 - 60 mL/min, lenalidomide dose determined in phase I, dexamethasone 40 mg orally days 1, 8, 15 and 22 of a 28 day cycle, and anticoagulants.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Anticoagulants
- Group B, CrCl < 30 mL/min (Experimental): Creatinine clearance < 30 mL/min, not on dialysis, lenalidomide dose determined in phase I, dexamethasone 40 mg orally days 1, 8, 15 and 22 of a 28 day cycle, and anticoagulants.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Anticoagulants
- Group C, CrCl < 30 mL/min, on dialysis (Experimental): Creatinine clearance < 30 mL/min and on dialysis, lenalidomide dose determined in phase I, dexamethasone 40 mg orally days 1, 8, 15 and 22 of a 28 day cycle, and anticoagulants.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Anticoagulants

INTERVENTIONS:
Drug: Lenalidomide — Given by mouth days 1-21 of a 28-day cycle. There is a 7 day rest (days 22-28). Continue until disease progression or unacceptable toxicity.
  Other Names: Revlimid
Drug: Dexamethasone — 40 mg given by mouth days 1, 8, 15 and 22 of a 28-day cycle. Continue until disease progression or unacceptable toxicity.
  Other Names: Decadron
Drug: Anticoagulants — Anticoagulation consisted of aspirin at either 81 mg/day or 325 mg/day at the physician's discretion. Heparin, low molecular weight heparin, or coumadin could be used if the patient was intolerant to aspirin.
  Other Names: Aspirin; Heparin; Low Molecular Weight Heparin; Coumadin

SUMMARY:
Patients with previously treated multiple myeloma and kidney dysfunction will be treated with lenalidomide and low-dose dexamethasone. Phase I will study the side effects and best dose of lenalidomide when given together with low-dose dexamethasone therapy. After the maximum safe and tolerated dose is found in Phase I, the study will proceed to Phase II. Phase II will study how well the the treatment works in patients with previously treated (relapsed or refractory) multiple myeloma and kidney dysfunction.

Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving lenalidomide together with dexamethasone may kill more cancer cells. Lenalidomide and dexamethasone may have different effects in patients who have changes in their kidney function.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) affects approximately 20,000 Americans annually and remains an incurable hematologic malignancy characterized by frequent early response followed by universal treatment relapse necessitating multiple sequential therapeutic regimens. Until recently, few effective therapies existed. Several novel agents for MM have now become available including the immunomodulatory drugs thalidomide, lenalidomide, as well as the proteasome inhibitor, bortezomib. Each of these agents is undergoing extensive clinical evaluation in combination with other therapies to produce unprecedented response rates in newly diagnosed and relapsed MM. Lenalidomide has proven to be a highly effective treatment agent, particularly when used in combination with dexamethasone but is renally excreted and little information is available about its use in myeloma patients with impaired kidney function (20% have renal failure at some time after diagnosis). Defining a safe and effective dose of lenalidomide to use is a critical step in MM treatment.

OUTLINE: This is a Phase I, dose-escalation study of lenalidomide followed by a Phase II study. Patients are stratified according to degree of renal dysfunction (moderate [creatinine clearance 30-60 mL/min] vs severe [creatinine clearance <30 mL/min and does not require dialysis] vs end-stage renal disease [creatinine clearance <30 mL/min and requires dialysis]).

Patients receive oral lenalidomide on days 1-21 and low-dose oral dexamethasone 40 mg on days 1, 8, 15, and 22. There is a 7 day rest (days 22-28) from lenalidomide. Each cycle is 28 days and repeated in the absence of disease progression or unacceptable toxicity.

Patients enrolled in the phase II portion of the study will undergo blood sample collection periodically for pharmacokinetic analysis of lenalidomide (Mayo Clinic sites only).

After completion of study treatment, patients are followed every 6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with previously treated multiple myeloma.
* Measurable disease assessed by one of the following ≤21 days prior to registration:

  * Serum monoclonal protein ≥1 g by protein electrophoresis
  * Urine monoclonal protein >200 mg on 24 hour electrophoresis
  * Serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis ≥30% (evaluable disease)
  * If both serum and urine m-components are present, both must be followed in order to evaluate response.
* All previous cancer therapy including chemotherapy, radiation, hormonal therapy and surgery, must be discontinued ≥2 weeks prior to registration.
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Acceptable organ and marrow function ≤21 days prior to registration:

  * Absolute neutrophil count (ANC) ≥1000/mm³
  * Platelet count ≥75,000/mm³
  * Total bilirubin ≤2 mg/dL
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 x upper limit of normal
* Renal impairment at baseline as measured by serum creatinine clearance (CrCl) ≤60 mL/min ≤21 days prior to registration.
* Females of Childbearing Potential (FCBP) must have a negative pregnancy test within 10-14 days and again within 24 hours of starting Cycle 1 and must use an effective double-method contraception for ≥28 days prior to, during, and for ≥28 days after completion of study therapy.
* Able to take required prophylactic anticoagulation.
* Able to understand and willingness to sign a written informed consent.
* Willing to provide blood samples for research purposes (Mayo Clinic sites only).
* If previously received lenalidomide, demonstration of clinical response of any duration or stable disease with progression-free interval of ≥6 months from start of that therapy.

Exclusion Criteria:

* Concurrent use of other anti-cancer agents or treatments. Growth factors and bisphosphonates are allowed as medically indicated. Steroids may be used with an equivalency of up to 20 mg of Prednisone per day as long as the dose has not been adjusted upwards in past 2 weeks prior to study registration.
* Uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection requiring IV antibiotics
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Uncontrolled cardiac arrhythmia
  * Psychiatric illness/social situation that would limit compliance with study requirements.
* Any of the following as this regimen may be harmful to a developing fetus or nursing child:

  * Pregnant women
  * Breast-feeding women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception.
* HIV-positive patients on combination antiretroviral therapy.
* Known hypersensitivity to thalidomide or other immunomodulatory drugs.
* History of Stevens-Johnson syndrome characterized by a desquamating rash while taking thalidomide or similar drugs.
* Other active malignancy except for non melanoma skin cancer or in situ cervical or breast cancer.
* Concurrent radiation therapy, except for palliation of a single painful bone lesion or fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-01-21 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2018-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R. Mikhael, MD, Study Chair — Mayo Clinic
Locations (16):
- United States (16):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Emory University Winship Cancer, Atlanta, Georgia
  - University of IL at Chicago, Chicago, Illinois
  - McFarland Clinic, Ames, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Michigan Cancer Research Consortium and Oncology Research- St. Joseph Mercy Hospital - Ann Arbor, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Metro MN CCOP, Saint Louis Park, Minnesota
  - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Kinston Medical Specialists, Kinston, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Reading Hospital and Medical Center, West Reading, Pennsylvania
  - WVU Mary Babb Randolph Cancer Center, Morgantown, West Virginia
  - Gundersen Lutheran, La Crosse, Wisconsin
  - Waukesha Memorial Hospital (ProHealth Care), Waukesha, Wisconsin
  - Aurora Cancer Center, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No
Data is proprietary.

REFERENCES:
- [Result] Mikhael J, Manola J, Dueck AC, Hayman S, Oettel K, Kanate AS, Lonial S, Rajkumar SV. Lenalidomide and dexamethasone in patients with relapsed multiple myeloma and impaired renal function: PrE1003, a PrECOG study. Blood Cancer J. 2018 Aug 29;8(9):86. doi: 10.1038/s41408-018-0110-7. PMID 30190454

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A Lenalidomide 10 mg/Day: Creatinine clearance (CrCl) of 30 - 60 mL/min. Lenalidomide 10 mg/day on days 1-21 and dexamethasone 40 mg/day on days 1, 8, 15 and 22 of a 28-day cycle. Anticoagulation consisting of aspirin at 81 or 325 mg/day at physician's discretion. Heparin, low molecular weight heparin, or coumadin could be used if the patient was intolerant to aspirin.
- Group A Lenalidomide 15 mg/Day: Creatinine clearance of 30 - 60 mL/min. Treated with lenalidomide 15 mg/day on days 1-21 and dexamethasone 40 mg/day on days 1, 8, 15 and 22 of a 28-day cycle. Anticoagulation consisting of aspirin at 81 or 325 mg/day at physician's discretion. Heparin, low molecular weight heparin, or coumadin could be used if the patient was intolerant to aspirin.
- Group A Lenalidomide 25 mg/Day: Creatinine clearance of 30 - 60 mL/min. Treated with lenalidomide 25 mg/day on days 1-21 and dexamethasone 40 mg/day on days 1, 8, 15 and 22 of a 28-day cycle. Anticoagulation consisting of aspirin at 81 or 325 mg/day at physician's discretion. Heparin, low molecular weight heparin, or coumadin could be used if the patient was intolerant to aspirin.
- Group B Lenalidomide 15 mg/2 Days: Creatinine clearance < 30 mL/min, not on dialysis. Treated with lenalidomide 15 mg/every other day on days 1-21 and dexamethasone 40 mg/day on days 1, 8, 15 and 22 of a 28-day cycle. Anticoagulation consisting of aspirin at 81 or 325 mg/day at physician's discretion. Heparin, low molecular weight heparin, or coumadin could be used if the patient was intolerant to aspirin.
- Group B Lenalidomide 25 mg/2 Days: Creatinine clearance of <30 mL/min, not on dialysis. Treated with lenalidomide 25 mg every other day for days 1-21 and dexamethasone 40 mg/day on days 1, 8, 15 and 22 of a 28-day cycle. Anticoagulation consisting of aspirin at 81 or 325 mg/day at physician's discretion. Heparin, low molecular weight heparin, or coumadin could be used if the patient was intolerant to aspirin.
- Group B Lenalidomide 15 mg/Day: Creatinine clearance < 30 mL/min, not on dialysis. Treated with lenalidomide at 15 mg/day for days 1-21 and dexamethasone 40 mg/day on days 1, 8, 15 and 22 of a 28-day cycle. Anticoagulation consisting of aspirin at 81 or 325 mg/day at physician's discretion. Heparin, low molecular weight heparin, or coumadin could be used if the patient was intolerant to aspirin.
- Group B Lenalidomide 25 mg/Day: Creatinine clearance < 30 mL/min, not on dialysis. Treated with lenalidomide at 25 mg/day for days 1-21 and dexamethasone 40 mg/day on days 1, 8, 15 and 22 of a 28-day cycle. Anticoagulation consisting of aspirin at 81 or 325 mg/day at physician's discretion. Heparin, low molecular weight heparin, or coumadin could be used if the patient was intolerant to aspirin.
- Group C Lenalidomide 15 mg 3x/Week: Creatinine clearance of 30 - 60 mL/min and on dialysis. Treated with lenalidomide 15 mg 3 days/week for days 1-21 and dexamethasone 40 mg/day on days 1, 8, 15 and 22 of a 28-day cycle. Anticoagulation consisting of aspirin at 81 or 325 mg/day at physician's discretion. Heparin, low molecular weight heparin, or coumadin could be used if the patient was intolerant to aspirin.
  Dialysis includes hemodialysis or peritoneal dialysis. When lenalidomide and/or dexamethasone treatment occurs on a dialysis day, lenalidomide and/or dexamethasone must be taken after dialysis.
- Group C Lenalidomide 10 mg/Day: Creatinine Clearance < 30 mL/min and on dialysis, treated with lenalidomide 15 mg 3 times per week, dexamethasone and anticoagulant
- Group C Lenalidomide 15 mg/Day: Creatinine Clearance < 30 mL/min and on dialysis, treated with lenalidomide 10 mg/day, dexamethasone, and anticoagulants
- Group C, Lenalidomide 25 mg/Day: Creatinine clearance < 30 mL/min and on dialysis, treated with lenalidomide at 25 mg/day, dexamethasone, and anticoagulants
Period: Dose Level 1
Arm/Group | Group A Lenalidomide 10 mg/Day | Group A Lenalidomide 15 mg/Day | Group A Lenalidomide 25 mg/Day | Group B Lenalidomide 15 mg/2 Days | Group B Lenalidomide 25 mg/2 Days | Group B Lenalidomide 15 mg/Day | Group B Lenalidomide 25 mg/Day | Group C Lenalidomide 15 mg 3x/Week | Group C Lenalidomide 10 mg/Day | Group C Lenalidomide 15 mg/Day | Group C, Lenalidomide 25 mg/Day
Started | 6 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Began Treatment | 6 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Completed (Treated until disease progression) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not Completed | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 2
Arm/Group | Group A Lenalidomide 10 mg/Day | Group A Lenalidomide 15 mg/Day | Group A Lenalidomide 25 mg/Day | Group B Lenalidomide 15 mg/2 Days | Group B Lenalidomide 25 mg/2 Days | Group B Lenalidomide 15 mg/Day | Group B Lenalidomide 25 mg/Day | Group C Lenalidomide 15 mg 3x/Week | Group C Lenalidomide 10 mg/Day | Group C Lenalidomide 15 mg/Day | Group C, Lenalidomide 25 mg/Day
Started | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 0 | 0
Began Treatment | 0 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Not Completed | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Intercurrent Illness/Other Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Period: Dose Level 3
Arm/Group | Group A Lenalidomide 10 mg/Day | Group A Lenalidomide 15 mg/Day | Group A Lenalidomide 25 mg/Day | Group B Lenalidomide 15 mg/2 Days | Group B Lenalidomide 25 mg/2 Days | Group B Lenalidomide 15 mg/Day | Group B Lenalidomide 25 mg/Day | Group C Lenalidomide 15 mg 3x/Week | Group C Lenalidomide 10 mg/Day | Group C Lenalidomide 15 mg/Day | Group C, Lenalidomide 25 mg/Day
Started | 0 | 0 | 7 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 0
Began Treatment | 0 | 0 | 6 | 0 | 0 | 3 | 0 | 0 | 0 | 3 | 0
Completed | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Not Completed | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Intercurrent Illness/Alternative Therapy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Ineligible/Withdrew before Treatment | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level 4
Arm/Group | Group A Lenalidomide 10 mg/Day | Group A Lenalidomide 15 mg/Day | Group A Lenalidomide 25 mg/Day | Group B Lenalidomide 15 mg/2 Days | Group B Lenalidomide 25 mg/2 Days | Group B Lenalidomide 15 mg/Day | Group B Lenalidomide 25 mg/Day | Group C Lenalidomide 15 mg 3x/Week | Group C Lenalidomide 10 mg/Day | Group C Lenalidomide 15 mg/Day | Group C, Lenalidomide 25 mg/Day
Started | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 5
Began Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0 | 0 | 0 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Period: Expansion Cohort
Arm/Group | Group A Lenalidomide 10 mg/Day | Group A Lenalidomide 15 mg/Day | Group A Lenalidomide 25 mg/Day | Group B Lenalidomide 15 mg/2 Days | Group B Lenalidomide 25 mg/2 Days | Group B Lenalidomide 15 mg/Day | Group B Lenalidomide 25 mg/Day | Group C Lenalidomide 15 mg 3x/Week | Group C Lenalidomide 10 mg/Day | Group C Lenalidomide 15 mg/Day | Group C, Lenalidomide 25 mg/Day
Started | 0 | 0 | 14 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Began Treatment | 0 | 0 | 14 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 7 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Closure | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible, treated patients
Groups:
- Group A=30-60 CrCl (mL/Min): Lenalidomide days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days. Phase I will determine the dose of lenalidomide to be used in Phase II.
  Group A=30-60 CrCl (mL/min): Each Cycle=28 days. Lenalidomide by mouth days 1-21 and Dexamethasone 40 mg by mouth days 1, 8, 15 and 22. There is a 7 day rest (days 22-28) from lenalidomide. Continue until disease progression or unacceptable toxicity. Phase I will determine the dose of lenalidomide to be used in Phase II.
- Group B=CrCL<30 mL/Min Not on Dialysis: Lenalidomide days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days. Phase I will determine the dose of lenalidomide to be used in Phase II.
  Group B=CrCL<30 mL/min not on dialysis: Each Cycle=28 days. Lenalidomide by mouth days 1-21 and Dexamethasone 40 mg by mouth days 1, 8, 15 and 22. There is a 7 day rest (days 22-28) from lenalidomide. Continue until disease progression or unacceptable toxicity. Phase I will determine the dose of lenalidomide to be used in Phase II.
- Group C=CrCL<30 mL/Min and on Dialysis: Lenalidomide days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days. Phase I will determine the dose of lenalidomide to be used in Phase II.
  Group C=CrCL<30 mL/min and on dialysis: Each Cycle=28 days. Lenalidomide by mouth days 1-21 and Dexamethasone 40 mg by mouth days 1, 8, 15 and 22. There is a 7 day rest (days 22-28) from lenalidomide. Continue until disease progression or unacceptable toxicity. Phase I will determine the dose of lenalidomide to be used in Phase II.
  Dialysis includes hemodialysis or peritoneal dialysis. When lenalidomide and/or dexamethasone treatment occurs on a dialysis day, lenalidomide and/or dexamethasone must be taken after dialysis.
- Total: Total of all reporting groups
Arm/Group | Group A=30-60 CrCl (mL/Min) | Group B=CrCL<30 mL/Min Not on Dialysis | Group C=CrCL<30 mL/Min and on Dialysis | Total
Number analyzed (Participants) | 29 | 19 | 14 | 62
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 73 [68 to 78] | 72 [62 to 79] | 64 [57 to 70] | 71.5 [64 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 6 | 31
  Male | 16 | 7 | 8 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 18 | 14 | 61
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 2 | 3 | 8
  White | 26 | 16 | 10 | 52
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Creatinine Clearance [Median (Inter-Quartile Range); unit: mL/min] — Serum creatinine clearance, mL/minute
  mL/min | 42.6 [37.0 to 51.2] | 22.8 [15.7 to 25.4] | 11.5 [9.7 to 17.2] | 27.4 [15.7 to 42.1]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Phase I Component With Dose Limiting Toxicities During the First Cycle of Therapy
Description: Dose Limiting Toxicity (DLT) was defined as any of the following events determined by the investigator to be possibly, probably, or definitely related to lenalidomide within the first cycle of therapy irrespective of whether the adverse events resolved:
  * Grade 3 or higher neutropenia with fever ≥38.5 degrees C
  * Grade 4 neutropenia ≥7 days
  * Grade 4 or higher thrombocytopenia
  * Other non-hematologic Grade 4 or higher adverse event not present prior to starting therapy or not due to underlying cause
Time Frame: First cycle of therapy (28 days)
Population: Patients treated during the dose finding phase of the study
Measure: Count of Participants; unit: Participants
Groups:
- Group A Lenalidomide 10 mg/Day: CrCl 30-60 mL/min, Lenalidomide at 10 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days along with anticoagulants.
- Group A Lenalidomide 15 mg/Day: CrCl 30-60 mL/min, Lenalidomide at 15 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days, along with anticoagulants.
- Group A Lenalidomide 25 mg/Day: CrCL 30-60 mL/min, Lenalidomide at 25 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days, along with anticoagulants.
- Group B Lenalidomide 15 mg/2 Days: CrCl<30 mL/min, not on dialysis, Lenalidomide at 15 mg/every 2 days for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days, along with anticoagulants.
- Group B Lenalidomide 25 mg/2 Days: CrCl < 30 mL/min, not on dialysis, Lenalidomide at 25 mg every 2 days for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days, along with anticoagulants.
- Group B Lenalidomide 15 mg/Day: CrCl < 30 mL/min, not on dialysis, Lenalidomide at 15 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days, along with anticoagulants.
- Group B Lenalidomide 25 mg/Day: CrCl < 30 mL/min, not on dialysis, Lenalidomide at 25 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days, along with anticoagulants.
- Group C Lenalidomide 15 mg 3x/Week: CrCl < 30 mL/min, on dialysis, Lenalidomide at 15 mg 3 times per week for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days, along with anticoagulants.
- Group C Lenalidomide 10 mg/Day: CrCl < 30 mL/min, on dialysis, Lenalidomide at 10 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days, along with anticoagulants.
- Group C Lenalidomide 15 mg/Day: CrCl < 30 mL/min, on dialysis, Lenalidomide at 15 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days, along with anticoagulants.
- Group C Lenalidomide 25 mg/Day: CrCl < 30 ml/min, on dialysis, Lenalidomide at 25 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days, along with anticoagulants.
Arm/Group | Group A Lenalidomide 10 mg/Day | Group A Lenalidomide 15 mg/Day | Group A Lenalidomide 25 mg/Day | Group B Lenalidomide 15 mg/2 Days | Group B Lenalidomide 25 mg/2 Days | Group B Lenalidomide 15 mg/Day | Group B Lenalidomide 25 mg/Day | Group C Lenalidomide 15 mg 3x/Week | Group C Lenalidomide 10 mg/Day | Group C Lenalidomide 15 mg/Day | Group C Lenalidomide 25 mg/Day
Number analyzed (Participants) | 6 | 3 | 6 | 3 | 3 | 3 | 8 | 3 | 3 | 3 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: Group A Lenalidomide 10 mg/Day vs Group A Lenalidomide 15 mg/Day vs Group A Lenalidomide 25 mg/Day; Recommended Phase 2 dose for Group A; Test type: Other — Recommended Phase 2 dose for Group A; Dose in milligrams per day = 25 — Because no dose limiting toxicities were noted, the recommended phase 2 dose for patients with creatinine clearance of 30 to 60 mL/min is 25 mg/day
Statistical Analysis 2: Comparison: Group B Lenalidomide 15 mg/2 Days vs Group B Lenalidomide 25 mg/2 Days vs Group B Lenalidomide 15 mg/Day vs Group B Lenalidomide 25 mg/Day; Recommended phase 2 dose for patients in Group B; Test type: Other — Recommended phase 2 dose for patients in Group B; Dose in milligrams/day = 25 — Because no dose limiting toxicities were noted, the recommended phase 2 dose of lenalidomide is 25 mg/day for patients with creatinine clearance < 30 mL/minute who are not on dialysis
Statistical Analysis 3: Comparison: Group C Lenalidomide 15 mg 3x/Week vs Group C Lenalidomide 10 mg/Day vs Group C Lenalidomide 15 mg/Day vs Group C Lenalidomide 25 mg/Day; Recommended phase 2 dose for Group C; Test type: Other — Recommended phase 2 dose for Group C; Lenalidomide dose in mg/day = 25 — Because no dose limiting toxicities were observed, the recommended phase 2 dose of lenalidomide is 25 mg/day for patients with creatinine clearance < 30 mL/min who are receiving dialysis

2. Primary Outcome: Percentage of Participants Who Experience a Response [sCR, CR, VGPR, PR]
Description: Per International Myeloma Working Group criteria, complete response (CR): negative immunofixation of serum and urine, normalization of free light chain (FLC) ratio if at study entry FLC was only measurable non-bone parameter, <5% plasma cells in bone marrow, disappearance of any soft tissue plasma cytomas; stringent complete response (sCR): all of above, + normal serum FLC ratio in all patients and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; partial response (PR): >=50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by >=90% or to < 200 mg per 24 hours, >=50% decrease in difference between involved and uninvolved FLC levels or a 50% decrease in level of involved FLC with 50% decrease in ratio, >=50% reduction in bone marrow plasma cells, if baseline percentage was >=30%, >=50% reduction in size of soft tissue plasmacytoma; very good partial response (VGPR): PR + improvements in serum and urine M-components
Time Frame: 56 months
Population: Patients treated at the recommended phase II dose
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Group A CrCl 30-60 mL/Min; Group B CrCL<30 mL/Min, Not on Dialysis: Lenalidomide at 25 mg/day days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group C CrCL<30 mL/Min and on Dialysis: Lenalidomide at 25 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
Arm/Group | Group A CrCl 30-60 mL/Min | Group B CrCL<30 mL/Min, Not on Dialysis | Group C CrCL<30 mL/Min and on Dialysis
Number analyzed (Participants) | 20 | 10 | 5
percentage of participants | 60.0 [39.4 to 78.3] | 60.0 [30.4 to 85.0] | 20.0 [1.0 to 65.7]

3. Secondary Outcome: Overall Survival Time
Description: Overall survival is the time from registration to death from any cause. Patients alive at the time of analysis were censored at the date last known alive.
Time Frame: 56 months
Population: Eligible, treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Group A=30-60 CrCl (mL/Min) | Group B=CrCL<30 mL/Min Not on Dialysis | Group C=CrCL<30 mL/Min and on Dialysis
Number analyzed (Participants) | 29 | 19 | 14
months | 20.8 [11.0 to 42.1] | 20.0 [10.4 to 34.2] | NA [10.4 to NA] — Insufficient observations to estimate median or upper confidence limit

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as time between the onset of response and disease progression in months, among patients treated at the recommended phase II dose who experienced a response to treatment. Per criteria of the International Myeloma Working Group, progressive disease was defined as one of the following: increase of 25% from best confirmed response in serum M-component, urine M-component, free light chain (FLC), bone marrow plasma cell percentage, or development of new or increase in size of bone lesions or soft tissue plasma cytomas. Development of hypercalcemia that can be attributed solely to the myeloma also constituted progression.
Time Frame: 56 months
Population: Patients treated at the recommended phase II dose who experienced a response to treatment
Measure: Median (Inter-Quartile Range); unit: Months
Groups:
- Group A=30-60 CrCl (mL/Min); Group B=CrCL<30 mL/Min Not on Dialysis: Lenalidomide 25 mg/day days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group C=CrCL<30 mL/Min and on Dialysis: Lenalidomide 25 mg/day days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days. Dialysis includes hemodialysis or peritoneal dialysis. When lenalidomide and/or dexamethasone treatment occurs on a dialysis day, lenalidomide and/or dexamethasone must be taken after dialysis.
Arm/Group | Group A=30-60 CrCl (mL/Min) | Group B=CrCL<30 mL/Min Not on Dialysis | Group C=CrCL<30 mL/Min and on Dialysis
Number analyzed (Participants) | 12 | 6 | 1
Months | 21.8 [14.4 to 34.8] | 8.4 [7.9 to 9.4] | 25.4 [25.4 to 25.4]

5. Secondary Outcome: Worst Degree Treatment-Related Adverse Events Across All Event Types Per Patient
Description: The highest degree of any adverse event experienced by each patient, as assessed by NCI CTCAE Version 4, with an attribution of possibly, probably, or definitely related to treatment. Reportable adverse events included those occurring while on treatment or within 30 days of the end of treatment.
Time Frame: 56 months
Population: All patients who started treatment
Measure: Number; unit: participants
Groups:
- Group A Lenalidomide 10 mg/Day: CrCl 30-60 mL/min, Lenalidomide 10 mg/day on days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group A Lenalidomide 15 mg/Day: CrCl 30-60 mL/min, Lenalidomide 15 mg/day on days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group A Lenalidomide 25 mg/Day: CrCl 30-60 mL/min, Lenalidomide 25 mg/day on days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group A Expansion Cohort: CrCl 30-60 mL/min, Lenalidomide 25 mg/day on days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days. Enrolled after determination of recommended phase 2 dose.
- Group B Lenalidomide 15 mg/2 Days: CrCl < 30 mL/min, not on dialysis. Lenalidomide days 15 mg every 2 days from days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group B Lenalidomide 25 mg/2 Days: CrCl < 30 mL/min, not on dialysis. Lenalidomide 25 mg every 2 days from days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group B Lenalidomide 15 mg/Day: CrCl < 30 mL/min, not on dialysis. Lenalidomide 15 mg/day on days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group B Lenalidomide 25 mg/Day: CrCl < 30 mL/min, not on dialysis. Lenalidomide 25 mg/day on days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group B Expansion Cohort: CrCl < 30 mL/min, not on dialysis. Lenalidomide 25 mg/day on days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days. Enrolled after determination of recommended phase 2 dose.
- Group C Lenalidomide 15 mg 3x/Week: CrCl < 30 mL/min, on dialysis, Lenalidomide 15 mg 3 times a week from days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group C Lenalidomide 10 mg/Day: CrCl < 30 mL/min, on dialysis, Lenalidomide 10 mg/day on days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group C Lenalidomide 15 mg/Day: CrCl < 30 mL/min, on dialysis, Lenalidomide 15 mg/day on days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group C Lenalidomide 25 mg/Day: CrCl < 30 mL/min, on dialysis, Lenalidomide 25 mg/day on days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
Arm/Group | Group A Lenalidomide 10 mg/Day | Group A Lenalidomide 15 mg/Day | Group A Lenalidomide 25 mg/Day | Group A Expansion Cohort | Group B Lenalidomide 15 mg/2 Days | Group B Lenalidomide 25 mg/2 Days | Group B Lenalidomide 15 mg/Day | Group B Lenalidomide 25 mg/Day | Group B Expansion Cohort | Group C Lenalidomide 15 mg 3x/Week | Group C Lenalidomide 10 mg/Day | Group C Lenalidomide 15 mg/Day | Group C Lenalidomide 25 mg/Day
Number analyzed (Participants) | 6 | 3 | 6 | 14 | 3 | 3 | 3 | 8 | 2 | 3 | 3 | 3 | 5
participants
  None | 3 | 1 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 0 | 2
  Grade 1 | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0
  Grade 2 | 2 | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
  Grade 3 | 1 | 1 | 4 | 6 | 1 | 1 | 1 | 3 | 0 | 0 | 1 | 1 | 3
  Grade 4 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

6. Secondary Outcome: Renal Function Over Time
Description: To describe renal function over time and to evaluate the safety profile of a onetime increase in lenalidomide dose at least 2 cycles after start of treatment due to improved renal function.
Time Frame: 56 months
Population: This outcome was not analyzed because the dose increase was not implemented.
Arm/Group | Group A=30-60 CrCl (mL/Min) | Group B=CrCL<30 mL/Min Not on Dialysis | Group C=CrCL<30 mL/Min and on Dialysis
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Pharmacokinetics of Lenalidomide in Impaired Renal Function
Description: To determine the pharmacokinetics of lenalidomide administration in myeloma patients with impaired renal function (pharmacokinetic analysis will be performed in up to 12 consented Mayo Clinic subjects treated during the Phase II component of the trial (only).
Time Frame: 56 months
Population: As only 1 patient was enrolled from Mayo Clinic during the Phase II component of the study, samples were neither collected nor analyzed for this endpoint.
Arm/Group | Group A=30-60 CrCl (mL/Min) | Group B=CrCL<30 mL/Min Not on Dialysis | Group C=CrCL<30 mL/Min and on Dialysis
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Progression-free Survival
Description: Progression-free survival is the time from registration to disease progression or death. Patients alive without disease progression were censored at the time of the last disease assessment.
Time Frame: 56 months
Population: Patients treated at the recommended phase II dose
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Group A=30-60 CrCl (mL/Min) | Group B=CrCL<30 mL/Min Not on Dialysis | Group C=CrCL<30 mL/Min and on Dialysis
Number analyzed (Participants) | 20 | 10 | 5
Months | 12.6 [6.5 to 25.1] | 11.4 [10.4 to 14.5] | NA [2.1 to NA] — Median and upper confidence limit are not estimable due to small sample size

ADVERSE EVENTS:
Time Frame: Adverse events were collected at every visit during treatment and for 30 days after the end of treatment (up to 56 months for at least 1 patient). The following events were captured: Grade 1 and 2 adverse events deemed possibly, probably or definitely related to study treatment; Grade 3 and 4 adverse events regardless of attribution, and any death within 30 days of the patient's last study treatment or procedure regardless of attribution.
Description: Serious adverse events include any adverse event occurring at least once at grade 3 or higher. The remaining adverse events occurring in at least 5% of patients (3 or more patients) are reported as other adverse events. Events were captured during each clinic visit while on treatment and for 30 days following the end of treatment.
Groups:
- Group A Lenalidomide 10 mg/Day: CrCl 30-60 mL/min. Lenalidomide 10 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group A Lenalidomide 15 mg/Day: CrCl 30-60 mL/min. Lenalidomide 15 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group A Lenalidomide 25 mg/Day: CrCl 30-60 mL/min. Lenalidomide 25 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group A Expansion Cohort: CrCl 30-60 mL/min. Lenalidomide 25 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days. Enrolled after determination of recommended phase 2 dose.
- Group B Lenalidomide 15 mg/2 Days: CrCl <30 mL/min, not on dialysis. Lenalidomide 15 mg every 2 days for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group B Lenalidomide 25 mg/2 Days: CrCl <30 mL/min, not on dialysis. Lenalidomide 25 mg every 2 days for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group B Lenalidomide 15 mg/Day: CrCl <30 mL/min, not on dialysis. Lenalidomide 15 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group B Lenalidomide 25 mg/Day: CrCl <30 mL/min, not on dialysis. Lenalidomide 25 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group B Expansion Cohort: CrCl <30 mL/min, not on dialysis. Lenalidomide 25 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days. Enrolled after determination of recommended phase 2 dose.
- Group C Lenalidomide 15 mg 3x/wk: CrCl < 30 mL/min, on dialysis. Lenalidomide 15 mg three times weekly for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group C Lenalidomide 10 mg/Day: CrCl < 30 mL/min, on dialysis. Lenalidomide 10 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group C Lenalidomide 15 mg/Day: CrCl < 30 mL/min, on dialysis. Lenalidomide 15 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
- Group C Lenalidomide 25 mg/Day: CrCl < 30 mL/min, on dialysis. Lenalidomide 25 mg/day for days 1-21 and Dexamethasone 40 mg days 1, 8, 15 and 22 every 28 days.
Arm/Group | Group A Lenalidomide 10 mg/Day | Group A Lenalidomide 15 mg/Day | Group A Lenalidomide 25 mg/Day | Group A Expansion Cohort | Group B Lenalidomide 15 mg/2 Days | Group B Lenalidomide 25 mg/2 Days | Group B Lenalidomide 15 mg/Day | Group B Lenalidomide 25 mg/Day | Group B Expansion Cohort | Group C Lenalidomide 15 mg 3x/wk | Group C Lenalidomide 10 mg/Day | Group C Lenalidomide 15 mg/Day | Group C Lenalidomide 25 mg/Day
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/3 | 0/6 | 4/14 | 0/3 | 0/3 | 0/3 | 0/8 | 0/2 | 0/3 | 1/3 | 1/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 5/6 | 2/3 | 5/6 | 10/14 | 3/3 | 3/3 | 1/3 | 5/8 | 1/2 | 2/3 | 3/3 | 3/3 | 4/5
Other Adverse Events (participants affected / at risk) | 5/6 | 2/3 | 6/6 | 14/14 | 1/3 | 3/3 | 3/3 | 8/8 | 2/2 | 1/3 | 2/3 | 3/3 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A Lenalidomide 10 mg/Day (N=6) | Group A Lenalidomide 15 mg/Day (N=3) | Group A Lenalidomide 25 mg/Day (N=6) | Group A Expansion Cohort (N=14) | Group B Lenalidomide 15 mg/2 Days (N=3) | Group B Lenalidomide 25 mg/2 Days (N=3) | Group B Lenalidomide 15 mg/Day (N=3) | Group B Lenalidomide 25 mg/Day (N=8) | Group B Expansion Cohort (N=2) | Group C Lenalidomide 15 mg 3x/wk (N=3) | Group C Lenalidomide 10 mg/Day (N=3) | Group C Lenalidomide 15 mg/Day (N=3) | Group C Lenalidomide 25 mg/Day (N=5)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Other (Eosinophilia) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Other (Pancytopenia) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other (Thrombocytopenia) (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Atrioventricular Block Complete (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Heart Failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous hemorrhage (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other (Diverticulitis) (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Death (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Other (Hepatic cirrhosis) (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other (Hepatobiliary disease) (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other (Cellulitis) (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other (Clostridial infection) (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other (Localized infection) (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Creatinine Increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
INR increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Other (pulmonary mass) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other (post-traumatic pain) (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Chronic kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other (Uremic encephalopathy) (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral ischemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thromboembolic Event (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A Lenalidomide 10 mg/Day (N=6) | Group A Lenalidomide 15 mg/Day (N=3) | Group A Lenalidomide 25 mg/Day (N=6) | Group A Expansion Cohort (N=14) | Group B Lenalidomide 15 mg/2 Days (N=3) | Group B Lenalidomide 25 mg/2 Days (N=3) | Group B Lenalidomide 15 mg/Day (N=3) | Group B Lenalidomide 25 mg/Day (N=8) | Group B Expansion Cohort (N=2) | Group C Lenalidomide 15 mg 3x/wk (N=3) | Group C Lenalidomide 10 mg/Day (N=3) | Group C Lenalidomide 15 mg/Day (N=3) | Group C Lenalidomide 25 mg/Day (N=5)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blurred vision (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Watering eyes (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other (Laceration) (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 4 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 3 | 3 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 6 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 5 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Other (Muscle spasms) (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 4 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 5 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2011-03-28): https://cdn.clinicaltrials.gov/large-docs/42/NCT00790842/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT00790842/SAP_001.pdf